CLINICAL TRIAL: NCT06026891
Title: Randomized, Double-blind, Placebo-controlled Phase III Clinical Study on the Effectiveness and Safety of MG-K10 Humanized Monoclonal Antibody Injection in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Study of MG-K10 Humanized Monoclonal Antibody Injection in Patients With Atopic Dermatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG-K10-AD-003
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Effectiveness of MG-K10 humanized monoclonal antibody injection in patients with moderate and severe atopic dermatitis Randomized, double-blind, placebo-controlled phase III clinical study with safety
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MG-K10 Humanized Monoclonal Antibody Injection (Experimental): Every four weeks, subcutaneous injection ，total of 52W
  Interventions: Drug: MG-K10/Placebo
- MG-K10 placebo (Placebo Comparator): Every four weeks, subcutaneous injection，The drug was transferred to the trial after 16 weeks
  Interventions: Drug: MG-K10/Placebo

INTERVENTIONS:
Drug: MG-K10/Placebo — MG-K10 Humanized Monoclonal Antibody Injection

SUMMARY:
The study is to reflect the effectiveness and safety of MG-K10 humanized monoclonal antibody injection in patients with moderate to severe atopic dermatitis.administered every 4 weeks for 52 week

DETAILED DESCRIPTION:
The study was a multicenter, randomized, double-blind, placebo-controlled Phase III study. Approximately 498 adults with moderate-to-severe AD who were not controlled by local therapy were scheduled to receive multiple subcutaneous injections (administered every 4 weeks for 52 weeks). The study was divided into screening period (1-5 weeks), double-blind treatment period (16 weeks), treatment maintenance period (36 weeks), and follow-up period (8 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years (inclusive of 18 and 75 years), both sexes;
2. patients with AD diagnosed in accordance with the American Academy of Dermatology Consensus Criteria (2014), with a pre-screening diagnosis of AD or history of eczema for ≥1 year, and the following:

   * Eczema Area and Severity Index (EASI) score ≥16 at screening and baseline visit;
   * Investigator's Overall Assessment (IGA) ≥3 points at screening and baseline visit;
   * BSA ≥10% of area of AD involvement at screening and baseline visit
   * Weekly mean of peak daily itch NRS score ≥4 at randomization;
3. the patient had an inadequate treatment effect on topical medication or systemic therapy within 6 months prior to the screening visit, or the use of topical medication or systemic therapy was medically inappropriate
4. negative screening blood pregnancy test results in women of childbearing age;

Exclusion Criteria.

1. subjects with a current diagnosis of other active skin disease (e.g., psoriasis or lupus erythematosus) that may interfere with AD evaluation;
2. Patients with ocular disease that, in the judgment of the Investigator, makes enrollment in the study inappropriate, e.g., past history of atopic keratoconjunctivitis with corneal involvement; if the Investigator is unable to make a determination, a diagnosis will be made by an ophthalmologist;
3. those who plan to undergo major surgery during the study period, including inpatient surgery and daytime outpatient surgery;
4. Subjects with the following conditions:

   * Persons who have used a biologic agent within 10 weeks prior to randomization or have not exceeded 5 half-lives (whichever is longer); Targeted inhibitors (e.g., JAK inhibitors, etc.), systemic glucocorticoids, cyclosporine and other immunosuppressants (e.g., methotrexate, mycophenolate mofetil [MMF], and azathioprine, etc.), phosphodiesterase (PDE4) inhibitors, ultraviolet light therapy, and systemic herbal medicine for AD within 4 weeks prior to randomization;
   * Has received topical glucocorticosteroids, topical calcineurin phosphatase inhibitors, antibiotic compound cream, and topical herbal therapy for AD within 1 week before randomization;
   * Has received allergen-specific immunotherapy within 6 months prior to randomization;
   * Live/live attenuated vaccination within 3 months prior to randomization or planned for the duration of the study;
   * Participation in a clinical study of another drug in the 3 months or 5 half-lives, whichever is longer, prior to randomization or planning to participate in a clinical study of another drug during the study period;
   * Subjects with prior use of an interleukin 4 receptor alpha subunit (IL-4Rα) monoclonal antibody drug who, in the judgment of the investigator, have developed drug resistance or drug-related serious AE;
   * Previous participation in the MG-K10 clinical trial;
5. evidence of active tuberculosis, or previous evidence of active tuberculosis without appropriate documented treatment; chest X-ray (frontal and lateral) or CT, etc. within 3 months prior to/surrounding the screening period suggesting the presence of active tuberculosis infection;
6. women who are breastfeeding or pregnant, or who plan to become pregnant or breastfeed during the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Estimated)
Dates: Start 2024-01-13 (Actual); Primary Completion 2025-06-11 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Proportions of subjects achieving EASI-75 | 16 weeks
  Proportions of subjects achieving EASI-75 (≥ 75% decrease from baseline in EASI
Proportions of subjects achieving IGA score of 0/1 point and a decrease of ≥ 2 | 16weeks
  Proportions of subjects achieving IGA score of 0/1 point and a decrease of ≥ 2 points from baseline

SECONDARY OUTCOMES:
The percentage of subjects who reached EASI-75 at other evaluation points; | 16 weeks
  The percentage of subjects who reached EASI-75 at other evaluation points;
Other evaluation points of view subjects with an IGA score of 0 or 1 | 16 weeks
  Other evaluation points of view subjects with an IGA score of 0 or 1 and a decrease of ≥ 2 points from the baseline
Percentage of subjects who reach EASI-50 | 16 weeks
  Percentage of subjects who reach EASI-50 (EASI score is ≥50% lower than the baseline)
Percentage of subjects who reach EASI-90 | 16 weeks
  Percentage of subjects who reach EASI-90 (EASI score is ≥90% lower than the baseline)
Each evaluation point of view EASI | 16 weeks
  Each evaluation point of view EASI score compared with the baseline change and change rate
Percentage of subjects with a decrease of ≥2 | 16 weeks
  Percentage of subjects with a decrease of ≥2 points from the baseline IGA score at each evaluation point of view
Percentage of subjects with a weekly average of daily peak itching NRS score ≥3 | 16 weeks
  Percentage of subjects with a weekly average of daily peak itching NRS score ≥3 points lower than the baseline;
The AD of each evaluation visit involves the change and rate of the baseline of BSA; | 16 weeks
  The AD of each evaluation visit involves the change and rate of the baseline of BSA;
The DLQI score of each evaluation interview has changed compared with the baseline. | 16 weeks
  The DLQI score of each evaluation interview has changed compared with the baseline.
The self-evaluation (POEM) score of patients with eczema from each evaluation point of view has changed compared with the baseline; | 16 weeks
  The self-evaluation (POEM) score of patients with eczema from each evaluation point of view has changed compared with the baseline;
The European Five-dimensional Health Scale (EQ-5D) | 16 weeks
  The European Five-dimensional Health Scale (EQ-5D) at each evaluation point of view is more than the baseline change and rate of change.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Medical Ph.D, Principal Investigator — Feking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No